CLINICAL TRIAL: NCT01766414
Title: In Vivo Effects of C1-esterase Inhibitor on the Innate Immune Response During Human Endotoxemia - A Randomized Controlled Pilot Study
Brief Title: In Vivo Effects of C1-esterase Inhibitor on the Innate Immune Response During Human Endotoxemia - VECTOR II
Acronym: VECTORII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 36688; 2011-002222-46 (EudraCT Number)
Record Dates: First submitted 2013-01-04; First posted 2013-01-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Innate Immune Response; Endotoxemia; Inflammation; Sepsis
MeSH Terms: conditions — Endotoxemia; Inflammation; Sepsis | interventions — Complement C1 Inhibitor Protein; let-363 protein, C elegans; Endotoxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C1-esterase inhibitor (Active Comparator): C1-esterase inhibitor 100 U/kg infusion followed by administration of Endotoxin 2ng/kg
  Interventions: Drug: C1-esterase inhibitor; Drug: Endotoxin
- Placebo (Placebo Comparator): Placebo (saline 0.9%) infusion followed by administration of Endotoxin 2ng/kg
  Interventions: Drug: Endotoxin

INTERVENTIONS:
Drug: C1-esterase inhibitor — intravenously
  Other Names: Cetor
  Arms: C1-esterase inhibitor
Drug: Endotoxin — intravenously
  Other Names: 2 ng/kg E. coli reference endotoxin 11:H 10:K negative

SUMMARY:
Excessive inflammation is associated with tissue damage caused by over-activation of the innate immune system. This can range from mild disease to extreme conditions, such as multiple organ dysfunction syndrome (MODS) and acute respiratory distress (ARDS). In marked contrast to adaptive immunity which is very sensitive to immune modulators such as steroids, the innate immune system cannot be sufficiently targeted by currently available anti-inflammatory drugs.

The investigators hypothesize that pre-treatment with C1-esterase inhibitor in a human endotoxemia model can modulate the innate immune response.

In this study, human endotoxemia will be used as a model for inflammation. Subjects will, prior to endotoxin administration, receive C1 esterase inhibitor or placebo. Blood will be sampled to determine the levels of markers of the innate immune response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers (18-35 years old)

Exclusion Criteria:

* Relevant medical history
* Drug-, nicotine-abuses
* Tendency towards fainting
* Hyper- or hypotension
* Use of any medication

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Neutrophil phenotype and redistribution | 8 hrs after LPS administration

SECONDARY OUTCOMES:
Cytokines and other markers of inflammation | 8 hrs after LPS administration
C1-inhibitor and complement concentration and activity | 8 hrs after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hoeven, Prof, Study Director — UMC Nijmegen
Locations (1):
- Radboud University, Nijmegen, Netherlands

REFERENCES:
- [Derived] Tak T, Wijten P, Heeres M, Pickkers P, Scholten A, Heck AJR, Vrisekoop N, Leenen LP, Borghans JAM, Tesselaar K, Koenderman L. Human CD62Ldim neutrophils identified as a separate subset by proteome profiling and in vivo pulse-chase labeling. Blood. 2017 Jun 29;129(26):3476-3485. doi: 10.1182/blood-2016-07-727669. Epub 2017 May 17. PMID 28515092